CLINICAL TRIAL: NCT01515007
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Pulmaquin® in the Management of Chronic Lung Infections With Pseudomonas Aeruginosa in Subjects With Non-Cystic Fibrosis Bronchiectasis, Including 28 Day Open-Label Extension and Pharmacokinetic Substudy (ORBIT-3)
Brief Title: Phase 3 Study With Ciprofloxacin Dispersion for Inhalation in Non-CF Bronchiectasis (ORBIT-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aradigm Corporation (Industry)
Collaborators: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Organization: Savara Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARD-3150-1201
Record Dates: First submitted 2012-01-10; First posted 2012-01-23 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Non Cystic Fibrosis Bronchiectasis
Keywords: Bronchiectasis, non-CF, Ciprofloxacin, Liposome
MeSH Terms: conditions — Bronchiectasis | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciprofloxacin dispersion for inhalation (Experimental): Liquid mixture of liposomally encapsulated and unencapsulated ciprofloxacin
  Interventions: Drug: Ciprofloxacin dispersion for inhalation
- Placebo (Placebo Comparator): Liquid formulation of empty liposomes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin dispersion for inhalation
  Other Names: Liquid mixture of liposomally encapsulated and unencapsulated ciprofloxacin
  Arms: Ciprofloxacin dispersion for inhalation
Drug: Placebo
  Other Names: Liquid formulation of empty liposomes
  Arms: Placebo

SUMMARY:
This study (ARD-3150-1201, ORBIT-3) will evaluate the safety and efficacy of inhaled Pulmaquin (ciprofloxacin dispersion for inhalation) compared to inhaled placebo in subjects who have a confirmed diagnosis of non-cystic fibrosis (non-CF) bronchiectasis with a history of pulmonary exacerbations and chronic P. aeruginosa infections.

ELIGIBILITY:
Inclusion Criteria:

* Verified bronchiectasis diagnosis
* Pseudomonas aeruginosa lung infection

Exclusion Criteria:

* Cystic Fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Time to first exacerbation | One Year

SECONDARY OUTCOMES:
Number of exacerbations | One Year

CONTACTS AND LOCATIONS:
Locations (109):
- United States (30):
  - Peoria, Arizona
  - Phoenix, Arizona
  - Downey, California
  - Los Angeles, California
  - Poway, California
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Celebration, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Sebring, Florida
  - Kailua, Hawaii
  - Chicago, Illinois
  - Columbia, Maryland
  - Royal Oak, Michigan
  - Rochester, Minnesota
  - Lincoln, Nebraska
  - Cedar Knolls, New Jersey
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Huntersville, North Carolina
  - Oklahoma City, Oklahoma
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Fort Worth, Texas
  - Tyler, Texas
  - Falls Church, Virginia
- Australia (9):
  - Concord, New South Wales
  - Westmead, New South Wales
  - Brisbane, Queensland
  - Cairns, Queensland
  - South Brisbane, Queensland
  - Daw Park, South Australia
  - Footscray, Victoria
  - Heidelberg, Victoria
  - Adelaide
- Canada (3):
  - Calgary, Alberta
  - Kelowna, British Columbia
  - Montreal, Quebec
- Germany (8):
  - Borstel, Schleswig-Holstein
  - Berlin
  - Donaustaff
  - Freiburg im Breisgau
  - Hanover
  - Immenstadt im Allgäu
  - Lübeck
  - Munich
- Hungary (4):
  - Budapest
  - Debrecen
  - Miskolc
  - Szombathely
- Ireland (2):
  - Dublin
  - Galway
- Israel (7):
  - Ashkelon
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Rehovot
  - Tel Aviv
- Italy (7):
  - Pavia, PV
  - Acquaviva delle Fonti
  - Bologna
  - Ferrara
  - Florence
  - Milan
  - Pisa
- Latvia (4):
  - Cekule
  - Daugavpils
  - Liepāja
  - Riga
- Poland (4):
  - Bialystok
  - Chrzanów
  - Warsaw
  - Wroclaw
- Romania (3):
  - Bucharest
  - Constanța
  - Timișoara
- South Africa (5):
  - Durban, KwaZulu-Natal
  - Pietermaritzburg, KwaZulu-Natal
  - Cape Town
  - eManzimtoti
  - Krugersdorp
- South Korea (2):
  - Busan
  - Seoul
- Spain (5):
  - Palma de Mallorca, Balearic Islands
  - Barcelona
  - Girona
  - Madrid
  - Málaga
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- United Kingdom (13):
  - Glasgow, Scotland
  - Birmingham, West Midlands
  - Bradford
  - Dundee
  - Liverpool
  - Llandough
  - London
  - Manchester
  - Newcastle upon Tyne
  - Nottinghamshire
  - Stoke-on-Trent
  - Tyne and Wear
  - Wolverhampton

REFERENCES:
- [Derived] Chalmers JD, Cipolla D, Thompson B, Davis AM, O'Donnell A, Tino G, Gonda I, Haworth C, Froehlich J. Changes in respiratory symptoms during 48-week treatment with ARD-3150 (inhaled liposomal ciprofloxacin) in bronchiectasis: results from the ORBIT-3 and -4 studies. Eur Respir J. 2020 Oct 22;56(4):2000110. doi: 10.1183/13993003.00110-2020. Print 2020 Oct. PMID 32554534
- [Derived] Haworth CS, Bilton D, Chalmers JD, Davis AM, Froehlich J, Gonda I, Thompson B, Wanner A, O'Donnell AE. Inhaled liposomal ciprofloxacin in patients with non-cystic fibrosis bronchiectasis and chronic lung infection with Pseudomonas aeruginosa (ORBIT-3 and ORBIT-4): two phase 3, randomised controlled trials. Lancet Respir Med. 2019 Mar;7(3):213-226. doi: 10.1016/S2213-2600(18)30427-2. Epub 2019 Jan 15. PMID 30658914